CLINICAL TRIAL: NCT05740891
Title: Clinical Study on the Safety and Effectiveness of Autologous Hematopoietic Stem Cell Transplantation Combined With CAR-T Cells in the Treatment of Refractory and Relapsed Multiple Myeloma
Brief Title: AHSCT Combined With CAR-T Cells in the Treatment of Refractory and Relapsed Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, The President of The First Affiliated Hospital, College of Medicine, Zhejiang University, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20210027C-R3
Record Dates: First submitted 2023-02-03; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma
Keywords: AHSCT; BCMA CAR-T
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Refractory and relapsed multiple myeloma
  Interventions: Drug: BCMA CAR-T cells injection

INTERVENTIONS:
Drug: BCMA CAR-T cells injection — Autologous hematopoietic stem cell transplantation combined with BCMA CAR-T cells

SUMMARY:
Clinical Study on the Safety and Effectiveness of Autologous Hematopoietic Stem Cell Transplantation Combined With CAR-T Cells in the Treatment of Refractory and Relapsed Multiple Myeloma

DETAILED DESCRIPTION:
This is a prospectiv , single arm, open-label, single-center study. This study is indicated for refractory and relapsed multiple myeloma. It aims to evaluate the safety and effectiveness of autologous hematopoietic stem cell transplantation combined with BCMA CAR-T to treat refractory and relapsed multiple myeloma. The main research is completely alleviated, overall reaction rate, and recurrence rate,etc. 50 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 1、BCMA positive accompanied by refractory/relapsed and resistance;
* 2、Patients with the tumor load is high and cannot be transplanted directly, before transplantation. Reduce the load through CAR-T treatment to prepare for transplantation;
* 3、Patient relapses after transplantation,donor lymphocyte infusion Invalid. The donor cells in the recipient body can be used or the donor cells can be collected directly.Prepare CAR-T to prevent recurrence and induce relapsing;
* 4、Repeated MRD (+) refractory drug resistant cases;
* 5、Male or female, 30-75 years old;
* 6、Anticipated survival time more than 12 weeks
* 7、Transplant subjects, regardless of their previous treatment, are eligible for inclusion after relapse；
* 8、Patients had a negative urine pregnancy test before the start of administration and agreed to take effective contraceptive measures during the test period until the last follow-up;
* 9、Those who voluntarily participate in the trial and sign the informed consent form

Exclusion Criteria:

* 1、Patients with the history of epilepsy or other CNS disease；
* 2、Patients with prolonged QT interval time or severe heart disease；
* 3、Pregnant or breastfeeding;
* 4、Active infection with no cure;
* 5、Patients with active hepatitis B or C infection;
* 6、Previously treated with any genetic therapy;
* 7、The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
* 8、Serum creatinine > 2.5mg/dl or ALT / AST > 3 times ULN or bilirubin > 2.0mg/dl;
* 9、Those who suffer from other uncontrolled diseases are not suitable to join the study;
* 10、HIV infection;
* 11、Any situation that the researchers believe may increase the risk of patients or interfere with the test results.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after BCMA CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | 24 months after cell infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
overall response rate | Up to 30 months
  The number of response patients/the number of total patients
Complete response rate(CRR) | Baseline up to 2 years after BCMA CAR T-cells infusion
  Proportion of subjects who achieved morphological complete response (CR) and complete response with hematologic incomplete recovery (CRi)
Overall survival (OS) | Month 6,12,18and 24
  Assessment of OS at Month 6,12,18and 24
Duration of response(DOR) | Month 6,12,18and 24
  Assessment of OS at Month 6,12,18and 24
Progression-free survival (PFS) | Month 6,12,18and 24
  Assessment of PFS at Month 6,12,18and 24

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China